CLINICAL TRIAL: NCT06020599
Title: Study of Pharmacological and Clinical Correlates of Frontal Cortical Electroencephalographic (EEG) Signal During the Induction, Maintenance and Emergence Phases of Anesthesia in Children
Acronym: SPECTRAL-PED
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230375
Record Dates: First submitted 2023-07-31; First posted 2023-08-31 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia
Keywords: anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children who need general anesthesia for surgery: Children who need general anesthesia for surgery (ENT, dentistry) at Louis Mourier Hospital.

SUMMARY:
Using data from a prospective cohort of children receiving general anaesthesia for surgery, this project will collect pharmacological correlates (doses and timing of administration of anaesthetic drugs) and clinical correlates (stimulations including nociceptive stimulation, possible responses such as movement/resumption of spontaneous ventilation during maintenance of anaesthesia/tachycardia/high blood pressure) of patients during the three phases of anesthesia (induction, maintenance, emergence).

DETAILED DESCRIPTION:
The usual practice of general anesthesia in children is based on the prescription of anesthetic drugs with doses adapted to weight and neurological examination focusing on the functions of the brainstem. Each patient has a specific sensitivity to anesthetic drugs (inter-individual pharmacokinetic and pharmacodynamic variability).

This inter-individual variability is likely to cause anesthesia that is too deep or, conversely, too light, which can be difficult to anticipate and can cause complications, particularly hemodynamic and neurocognitive. Because of the pharmacokinetics of anesthetic drugs, once an overdose is present, it will be relatively prolonged (several minutes). This is the correction of overdose.

In adults, monitoring of anesthesia adequacy is performed by EEG signal analysis (mainly BIS (Bispectral Index) monitor, Medtronic, Dublin, Ireland). This practice is not very common in children.

Since 2020, an EEG monitor (Sedline, Masimo, Irvine, California, USA) allows the estimation of the adequacy of anesthesia in children based on an EEG model (spectral density matrix; double spectrum delta and alpha during the maintenance phase of anesthesia).

Nevertheless, the pharmacological correlates (doses and delays in reaching the peak of the effect of drugs) as well as the clinical correlates (loss of verbal contact at induction, responses to nociceptive stimuli during the maintenance of anesthesia, return of brainstem functions in the emerging phase) associated with this double delta/alpha spectrum are not described. In addition, monitor EEG analysis tools cannot correctly describe (in spectral density matrix) the induction and emergence (awakening) phases of general anesthesia.

Questions remain about the potentially deleterious effects of general anesthesia in children, especially in children under one year of age. To the extent that general anesthesia is necessary for the performance of the surgical procedure, it is essential to have tools (cortical EEG) that make it possible to adjust the doses of anesthetic drugs to adapt to inter-individual variability. In children, the use of EEG for estimating the adequacy of anaesthesia remains incomplete and imperfect.

ELIGIBILITY:
Inclusion Criteria:

* 1 year < age < 18 years
* Weight> 10 kg
* Child receiving general anesthesia for any scheduled surgical procedure (dentistry and ENT) at Louis Mourier Hospital
* Information for holders of parental authority

Exclusion Criteria:

* Child with known autism disorder
* Refusal of parental authority holders to participate or refusal of the child
* Participation in other intervention research
* Not affiliated to a social security system

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children requiring general anesthesia for surgery (ENT, dentistry) at Louis Mourier Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Pharmacological correlates (doses and timing of administration of anaesthetic drugs) of patients during the three phases of anaesthesia (induction/maintenance/emergence). | 6 months
  The aim is to assert that a given EEG profile (described by the spectral density matrix, by the unique digital descriptors and by the analogue EEG) is associated with such doses/concentrations of drugs and is associated with probabilities of response (movement/haemodynamics).
Clinical correlates (stimulations including nociceptive stimulation, possible responses such as movement/resumption of spontaneous ventilation during maintenance of anaesthesia/tachycardia/hypertension) of patients during the three phases of anaesthesia. | 6 months
  The aim is to assert that a given EEG profile (described by the spectral density matrix, by the unique digital descriptors and by the analogue EEG) is associated with such doses/concentrations of drugs and is associated with probabilities of response (movement/haemodynamics).

SECONDARY OUTCOMES:
The calculation of the delta-alpha ratio to help the development of mathematical tools to quantify delta-alpha spectra images on the spectral density matrix during the maintenance phase of anesthesia | 6 months
Intra-individual correlation of sensitivity between the different phases of anesthesia (induction-maintenance-emergence) | 6 months
  This is to test the hypothesis that a patient identified as sensitive during the induction phase (time required to move from a delta trace with superimposed alpha to a trace with exclusive delta waves) will also be sensitive (will need lower doses/concentrations of hypnotics) to have a double delta-alpha spectrum during the maintenance phase of anesthesia. If this interindividual sensitivity persists, the patient will need to emerge from anesthesia (persistence of fast waves) at lower concentrations of hypnotics compared to less sensitive patients.
Sensitivity and specificity of a typical EEG profile (persistent beta/gamma waves) to help predicting extubation against currently used clinical and "scientific" criteria. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan Longrois, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Louis Mourier, Colombes, France

IPD SHARING:
Plan to Share IPD: No